CLINICAL TRIAL: NCT00118859
Title: Model of Integrative Care in an Academic Health Center
Brief Title: Pilot Study to Test the Effectiveness of Combining Conventional and Complementary Medicine to Treat Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AT000905 (NIH); ICC
Record Dates: First submitted 2005-07-07; First posted 2005-07-12 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Low Back Pain
Keywords: Back Pain; Integrative Care; Acupuncture; Chiropractic; Exercise; Massage Therapy; Mind-Body Therapy; Nutritional Counseling; Complementary Therapies; Complementary and Alternative Medicine
MeSH Terms: conditions — Low Back Pain; Back Pain; Motor Activity

INTERVENTIONS:
Behavioral: Integrative care for low back pain
Behavioral: Conventional treatment for low back pain

SUMMARY:
This pilot study will determine the feasibility of enrolling participants from different populations for a larger study of low back pain (LBP) treatment. In addition, this study will assess the effectiveness of data collection instruments and procedures as well as utilize feedback from participants to refine a future study.

DETAILED DESCRIPTION:
Back pain is one of the most common health problems in the United States, afflicting up to 50% of adults each year. Back pain is the leading cause of visits to orthopedic surgeons and the second leading cause of visits to general practitioners. In the United States, the estimated annual cost of back pain, including medical costs and lost productivity, is between $50 and $100 billion. Unfortunately, conventional medical care has been largely ineffective in treating back pain of most people. An increasing number of people with back pain, particularly with LBP, are seeking relief from unconventional sources such as chiropractors and massage therapies. Although complementary and alternative medicine (CAM) therapies are being used to treat LBP, their effectiveness has not been thoroughly examined. Even less is known about the effectiveness of combining conventional medical care with CAM therapies to provide "integrative care." This pilot study will recruit participants from three different patient populations to determine the effectiveness of integrative care in treating LBP symptoms.

This study will last 26 weeks and will comprise three participant populations: patients at an occupational health clinic, primary care patients at a medical clinic, and workers' compensation patients at the same medical clinic. At study start, participants will be interviewed about the care they have already received for LBP, any activities limited by their LBP, their attitudes toward CAM back pain treatments, job satisfaction, social support in the workplace, and medical history. Participants will also complete a self-report pain scale and a disability questionnaire. Participants will then be randomly assigned to either receive treatment for their LBP at an Integrative Care Center or continue to receive usual care provided by their medical or occupational health clinic.

Participants assigned to receive integrative care will be evaluated by both a medical doctor and a CAM clinician immediately after being interviewed. Following the evaluation, the two clinicians will meet and develop a treatment plan, which will include conventional medical care and some form of CAM such as acupuncture, chiropractic, exercise, massage, mind-body therapy, or nutritional counseling. Treatments will occur either once or twice weekly for the 12-week duration of treatment; clinicians may revise treatment plans during the study. LBP symptoms will be assessed through phone interviews at Weeks 2, 5, 12, and 26.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain beginning 3 to 6 weeks prior to study entry
* Patient of Partners Occupational Health Center or Harvard Vanguard Medical Associates (HVMA)
* Able to speak and understand English
* Willing and able to comply with all study requirements

Exclusion Criteria:

* History of back surgery within 3 years prior to study entry
* History of vertebral fracture or dislocation
* Progressive or severe neurological symptoms such as loss of bowel or bladder control, numbness in groin or rectal area, or extreme leg weakness
* Severe inflammation of the vertebrae, stiffening of the joints and ligaments, or scoliosis
* Pacemaker or implanted defibrillator
* Underlying systemic or visceral disease which might be causing back pain
* Osteoporosis
* Cancer within 5 years prior to study entry. Participants with non-melanoma skin cancer are not excluded.
* Unexplained weight loss or recent unexplained fever
* Bleeding disorder or current use of anticoagulant medication
* Any disabling medical condition
* Major organ transplantation
* Current use of systemic corticosteroids
* Current use of immunosuppressive medications
* Current use of intravenous drugs
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-07; Study Completion 2006-04

PRIMARY OUTCOMES:
LBP symptoms

SECONDARY OUTCOMES:
Feasibility of enrolling LBP patients from different populations
effectiveness of data collection instruments and procedures

CONTACTS AND LOCATIONS:
Overall Officials: David Eisenberg, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)